CLINICAL TRIAL: NCT00786370
Title: Dexmedetomidine vs. Propofol for Monitored Anesthesia Care During Cataract
Brief Title: Dexmedetomidine vs. Propofol for Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Jeffrey Littman, MD, Cooper University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 08-045
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2008-11

CONDITIONS: Cataract
Keywords: propofol; dexmedetomidine; cataract; respiratory; blood pressure; Cataract surgery
MeSH Terms: conditions — Cataract | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator)
  Interventions: Drug: Propofol
- Dexmedetomidine (Experimental)
  Interventions: Drug: dexmedetomidine; Drug: Dexemedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — Propofol or dexmedetomidine infusion will be started according to the randomized treatment allocation. The propofol group will receive a bolus of 2mg midazolam and 100mcg fentanyl and then continuous propofol infusion at 50-100mcg/kg/min until a Ramsay score of 3 or Bis score of 60-80 is achieved. The dexmedetomidine group will receive a bolus of dexmedetomidine 1mcg/kg for 10 minutes and then a continuous infusion of dexmedetomidine 0.2-0.7mcg/kg/hr until a Ramsay score of 3 or a Bis score of 60-80 are achieved.
  Arms: Dexmedetomidine
Drug: Propofol — continuous propofol infusion at 50-100mcg/kg/min until a Ramsay score of 3 or Bis score of 60-80 is achieved
  Arms: Propofol
Drug: Dexemedetomidine — continuous infusion of dexmedetomidine 0.2-0.7mcg/kg/hr until a Ramsay score of 3 or a Bis score of 60-80 are achieved.
  Arms: Dexmedetomidine

SUMMARY:
The use of dexmedetomidine in cataract surgery is still limited and to date only one study has examined anesthetic technique in this patient population. This pilot study will therefore compare the use of dexmedetomidine and propofol in subjects undergoing cataract surgery. The primary endpoint will be based on simple cardiorespiratory measures often associated with complications from sedation as well as assessment of the achieved sedation by the attending anesthesiologist and surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Normal renal function
2. No chronic use of narcotics
3. ASA PS1-3
4. Males or females age 18 or older

Exclusion Criteria:

1. Liver disease (Child Pugh classification 1-3)
2. History of chronic use of sedatives, narcotics, alcohol or illicit drugs or allergy to any the study medications
3. History of 1st and 2nd degree heart block (not paced)
4. Any patient with EF < 30%
5. Patients with active seizure history
6. Pregnant patients (women of child bearing potential will have a preoperative pregnancy test as is standard of practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To compare select cardiorespiratory effects of dexmedetomidine sedation to those of propofol sedation in patients undergoing cataract surgery. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Littman, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States